CLINICAL TRIAL: NCT04933812
Title: EngagINg the COmmunity to Reduce Preterm Birth Via Adherence To an Individualized Prematurity Prevention Plan (INCORPorATe IP3)
Brief Title: EngagINg the COmmunity to Reduce Preterm Birth Via Adherence To an Individualized Prematurity Prevention Plan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00107668
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Intervention Arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Social Support Meetings and Facebook Group (Other): Facebook group where community doulas will be providing information on various pregnancy and support topics in addition to 8 possible group Zoom meetings that will include pregnancy-related/reflection topics.
  Interventions: Behavioral: Facebook discussions and Virtual group meetings

INTERVENTIONS:
Behavioral: Facebook discussions and Virtual group meetings — Participants must join a study-specific private Facebook group and engage in discussion. Once the discussion is complete, participants have the opportunity to join virtual group sessions via Zoom

SUMMARY:
The purpose of this study is to determine if INCORPorATe IP3 is feasible prior to a larger trial focused on determining efficacy. Feasibility will be measured using the RE-AIM framework4: Reach or Participation (Primary Outcome): (a) percent of eligible participants who are successfully recruited and attend at least one group session; Effectiveness: retention rate in the intervention; Implementation: fidelity to the intervention protocol; Maintenance: intervention sustainability based on continued engagement from the participants.

DETAILED DESCRIPTION:
Non-Hispanic black (NHB) women are 49% more likely to experience a preterm birth (PTB), delivery before 37 weeks. PTB is associated with increased risk of poor short and long-term neonatal outcomes. PTB can occur in multiple clinical scenarios including spontaneous PTB (e.g. preterm labor, preterm pre-labor rupture of membranes) and medically induced preterm labor (e.g. preeclampsia). Women with a history of PTB are at 1.5 - 2 fold increased risk for future PTB. There are medical therapies than can reduce the risk of recurrent PTB specific to the presumed etiology of the prior PTB. Thus, women with a history of a prior PTB who receive care with Duke Maternal Fetal Medicine (MFM) receive and Individualized Prematurity Prevention Plan (IP3) to reduce their risk of recurrent PTB. The IP3 plans are often labor intensive with requirements ranging from daily medications, weekly clinic visits, painful injections or invasive ultrasounds.

Given the increased rate so of PTB among NHB women and some suggestion of decreased adherence in this population1, we previously conducted qualitative studies with NHB women to uncover patient perceived barriers to IP3 adherence2,3. These studies revealed that NHB women with prior preterm birth felt that stress and lack of support were key barriers to preterm birth prevention adherence. Stress and limited support made women feel isolated from their peers and community. Based on these data we worked with a stakeholder group to develop a patient-centered, community-involved intervention that will increased adherence to an individualized prematurity prevention plan using community-level social supports. The resulting invention titled, EngagINg the COmmunity to Reduce Preterm Birth via Adherence To an Individualized Prematurity Prevention Plan (INCORPorATe IP3) includes community doula led group social support.

ELIGIBILITY:
Inclusion Criteria:

* self describe race as Non-hispanic black
* history of prior singleton preterm delivery (before 37 weeks gestation
* current singleton gestation, with Individualized Prematurity Prevention (IP3) plan.

Exclusion Criteria:

* women with anomalous fetuses
* age below 18 years
* non-English speaking

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarahn Wheeler, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wheeler SM, Massengale KEC, Fitzgerald TA, Truong T, Ostbye T, Corneli A, Swamy GK. IMPaCT: A Pilot Randomized Trial of an Intervention to Reduce Preterm Birth Among Non-Hispanic Black Patients at High Risk. Health Equity. 2022 Dec 19;6(1):922-932. doi: 10.1089/heq.2022.0089. eCollection 2022. PMID 36636112

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group Social Support Meetings and Facebook Group
Started | 31
Completed | 29
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Arm/Group | Group Social Support Meetings and Facebook Group
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 29
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Eligible Participants Who Are Successfully Recruited and Attend at Least One Group Session
Time Frame: up to 12 weeks after delivery (approximately 1 year)
Measure: Count of Participants; unit: Participants
Arm/Group | Group Social Support Meetings and Facebook Group
Number analyzed (Participants) | 29
Participants | 20

2. Primary Outcome: Number of Sessions Attended by Each Participant
Description: As a measure of effectiveness
Time Frame: up to 12 weeks after delivery (approximately 1 year)
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Group Social Support Meetings and Facebook Group
Number analyzed (Participants) | 29
sessions | 5.7 (6.9)

3. Primary Outcome: Implementation as Measured by the Number of Sessions Including Each Topic
Time Frame: up to 12 weeks after delivery (approximately 1 year)
Measure: Count of Units; unit: Sessions
Units Other Than Participants: Sessions
Arm/Group | Group Social Support Meetings and Facebook Group
Number analyzed (Participants) | 29
Number analyzed (Sessions) | 51
Sessions
  Individualized Prematurity Prevention Plan | 14
  Changing Baby - Changing You | 31
  TEAMING UP Together | 14
  Preterm Labor - Warning Signs / Symptoms | 7
  The Labor Process | 13
  Pregnancy Progression | 5
  Late Pregnancy Warning Signs | 9
  Reunion | 5

4. Primary Outcome: Engagement as Measured by Number of Participants Who Attended More Than One Session
Description: Intervention sustainability based on continued engagement from the participants
Time Frame: up to 12 weeks after delivery (approximately 1 year)
Measure: Count of Participants; unit: Participants
Arm/Group | Group Social Support Meetings and Facebook Group
Number analyzed (Participants) | 29
Participants | 17

5. Primary Outcome: Engagement as Measured by Number of Participants Who Completed PSA (Pregnancy-specific Anxiety), IPC-18 (Interpersonal Processes of Care), MSSS (Maternal Social Support Scale), and CSQ-9 (Client Satisfaction Questionnaire) at All Time Points
Description: Intervention sustainability based on continued engagement from the participants
Time Frame: up to 12 weeks after delivery (approximately 1 year)
Measure: Count of Participants; unit: Participants
Arm/Group | Group Social Support Meetings and Facebook Group
Number analyzed (Participants) | 29
Participants | 22

6. Secondary Outcome: IP3 Knowledge Questionnaire
Description: Questionnaire includes approximately four questions aimed to evaluate a participants knowledge about the details of their IP3 plan. Participants will only receive questions that pertain to their specific IP3. They will be given the answers immediately following the assessment. Understanding of preterm birth and precautions; higher scores better, each questionnaire ranges from 0 to 5 questions correct
Time Frame: at intake
Population: Participants who received each question per their IP3 plan.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Social Support Meetings and Facebook Group
Number analyzed (Participants) | 29
score on a scale
  Cervix length and cerclage: number analyzed (Participants) | 16
  Cervix length and cerclage | 2.6 (0.6)
  Progesterone therapy: number analyzed (Participants) | 15
  Progesterone therapy | 2.3 (1.0)
  Low dose aspirin: number analyzed (Participants) | 20
  Low dose aspirin | 3.0 (0.9)
  Lifestyle modification | 3.1 (1.1)

7. Secondary Outcome: Pregnancy-specific Anxiety (PSA)
Description: The PSA is a validated 13-item tool used to assess anxiety specific to pregnancy this tool has been correlated with preterm birth outcome. On a Likert scale of 1 to 5, higher scores indicate greater anxiety.
Time Frame: At intake and at gestational age 20-28 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Social Support Meetings and Facebook Group
Number analyzed (Participants) | 29
score on a scale
  At intake | 2.7 (1.0)
  At Gestational Age 20-28 weeks | 2.2 (1.0)

8. Secondary Outcome: Interpersonal Processes of Care (IPC)
Description: The IPC is an 18-question questionnaire that asks participants about their experience with receiving care within a specific clinic (in this case the Duke Perinatal Durham Clinic). On a Likert scale of 1 to 5, higher scores indicate more of the item being measured.
Time Frame: at intake
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Social Support Meetings and Facebook Group
Number analyzed (Participants) | 29
score on a scale
  Lack of clarity | 1.9 (0.9)
  Elicited concerns, responded | 4.5 (0.6)
  Explained results | 4.7 (0.7)
  Decided together | 4.4 (0.7)
  Emotional support, compassion | 4.7 (0.6)
  Discriminated due to race/ethnicity | 1.2 (0.6)
  Disrespectful office staff | 1.1 (0.4)

9. Secondary Outcome: Interpersonal Processes of Care (IPC)
Description: as for outcome 8
Time Frame: Gestational age 20-28 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Social Support Meetings and Facebook Group
Number analyzed (Participants) | 29
score on a scale
  Lack of clarity | 1.4 (0.9)
  Elicited concerns, responded | 4.4 (0.8)
  Explained results | 4.6 (0.5)
  Decided together | 4.4 (0.7)
  Emotional support, compassion | 4.6 (0.6)
  Discriminated due to race/ethnicity | 1.4 (0.8)
  Disrespectful office staff | 1.3 (0.8)

10. Secondary Outcome: Interpersonal Processes of Care (IPC)
Description: as for outcome 8
Time Frame: Gestational age >= 30 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Social Support Meetings and Facebook Group
Number analyzed (Participants) | 29
score on a scale
  Lack of clarity | 1.8 (0.9)
  Elicited concerns, responded | 4.5 (0.6)
  Explained results | 4.6 (0.7)
  Decided together | 4.5 (0.7)
  Emotional support, compassion | 4.6 (0.8)
  Discriminated due to race/ethnicity | 1.4 (0.8)
  Disrespectful office staff | 1.1 (0.3)

11. Secondary Outcome: Maternal Social Support Scale (MSSS)
Description: The MSSS is a six-question scale that quantifies a pregnant women's social support as low, medium or adequate. On a Likert scale of 1 to 5, higher scores indicate greater social support.
Time Frame: At intake, gestational age 20-28 weeks, and gestational age >=30 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Social Support Meetings and Facebook Group
Number analyzed (Participants) | 29
score on a scale
  At intake | 27.3 (3.4)
  Gestational age 20-28 weeks | 28.2 (3.0)
  Gestational age >= 30 weeks | 27.7 (4.0)

12. Secondary Outcome: Number of Participants Who Were Adherent to the IP3 Plan
Description: Adherence to the IP3 based on both participant report and EHR chart review; dichotomized as adherent or not adherent.
Time Frame: Post delivery (up to approximately 40 weeks)
Population: Participants to which the measure was relevant.
Measure: Count of Participants; unit: Participants
Arm/Group | Group Social Support Meetings and Facebook Group
Number analyzed (Participants) | 29
Participants
  IOM weight gain guidelines: number analyzed (Participants) | 16
  IOM weight gain guidelines | 8
  Tobacco cessation: number analyzed (Participants) | 5
  Tobacco cessation | 2
  17-P: number analyzed (Participants) | 15
  17-P | 6
  Progesterone: number analyzed (Participants) | 1
  Progesterone | 0
  Cerclage: number analyzed (Participants) | 8
  Cerclage | 7
  Serial cervix length: number analyzed (Participants) | 13
  Serial cervix length | 6
  Low dose aspirin: number analyzed (Participants) | 28
  Low dose aspirin | 13

ADVERSE EVENTS:
Time Frame: Up to 12 weeks after delivery (approximately 1 year)
Arm/Group | Group Social Support Meetings and Facebook Group
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group Social Support Meetings and Facebook Group (N=31)
IUFD (Intrauterine Fetal Demise) (Pregnancy, puerperium and perinatal conditions) | 1 — Unrelated to study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT04933812/Prot_001.pdf
  • Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT04933812/SAP_002.pdf
  • Informed Consent Form (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT04933812/ICF_000.pdf